CLINICAL TRIAL: NCT06387407
Title: Population Pharmacokinetic Study of the Effect of Polymorphisms in the ABCB1 and CES1 Genes on the Pharmacokinetics of Dabigatran
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Yan He, Professor, The Affiliated Hospital Of Guizhou Medical University
Other Study IDs: 2024037K
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Combined Analysis of Polymorphisms and Dabigatran Pharmacokinetic Parameters
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dabigatran Etexilate 150mg — Oral dabigatran etexilate capsules, 150 mg twice a day.

SUMMARY:
According to published studies, the effects of genetic polymorphisms in the ABCB1 and CES1 genes on the blood concentration of dabigatran are controversial, and it is not clear whether dabigatran dosage and dosing intervals need to be adjusted according to genotype or other covariates in Chinese subjects. For these purposes, we will include patient demographics, genetic polymorphisms, and PK data based on a population pharmacokinetic study of dabigatran ester in healthy Chinese subjects to analyze the effect on dabigatran pharmacokinetics.

The aim of this study was to develop a population pharmacokinetic model to understand the relationship between dabigatran-related genes and dabigatran plasma levels after a single oral dose in healthy Chinese subjects and patients, and to analyze the effects of genetic variation on the efficacy and safety of dabigatran etexilate.

ELIGIBILITY:
Inclusion and exclusion criteria for healthy subjects were consistent with bioequivalence studies.

Inclusion Criteria:

1. Age 18-89 years;
2. ECG meeting the diagnostic criteria for atrial fibrillation;
3. Provide at least one valid blood sample for SNP testing;
4. no contraindication to anticoagulation, blood counts and coagulation times within normal reference values, and negative urine and stool occult blood;
5. not have had any stroke in the 6 months prior to enrollment.

Exclusion Criteria:

1. Cardiac ultrasound suggestive of moderate-to-severe mitral stenosis or after mechanical valve replacement;
2. severe hepatic injury or renal insufficiency (estimated glomerular filtration rate [eGFR] <30 mL/(min*1.73m2))
3. History of stroke or peripheral arterial embolism during dosing;
4. patients at high risk of bleeding, such as history of bleeding, hematologic disorders, other disorders requiring anticoagulant therapy, peptic ulcer and other bleeding, and blood pressure >180/110 mmHg;
5. Combination of other serious diseases, such as malignant tumors, severe hepatic and renal insufficiency;
6. history of allergy to dabigatran and warfarin.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects in the dabigatran etexilate bioequivalence study; patients with nonvalvular atrial fibrillation (NVAF).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentration | 3 day
  Blood samples collected 10-16 hours after the previous dose were considered trough plasma levels of dabigatran, and blood samples collected 1-3 hours after the dose were considered peak plasma levels.